CLINICAL TRIAL: NCT02365493
Title: CAMERA 2 - Combination Antibiotic Therapy for Methicillin Resistant Staphylococcus Aureus Infection - An Investigator-initiated, Multi-centre, Parallel Group, Open Labelled Randomised Controlled Trial
Brief Title: Combination Antibiotic Therapy for Methicillin Resistant Staphylococcus Aureus Infection
Acronym: CAMERA2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recommendation of the Data Safety Monitoring Committee
Sponsor: Menzies School of Health Research (Other)
Collaborators: Australasian Society for Infectious Diseases (Other); Singapore Infectious Diseases Clinical Research Network (Other); The University of Queensland (Other); Australasian Kidney Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHMRC1078930
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
Keywords: Methicillin-Resistant Staphylococcus aureus (MRSA)
MeSH Terms: interventions — beta-Lactams; Floxacillin; Cloxacillin; Cefazolin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard therapy (No Intervention): Intravenous vancomycin dosed as per Australian Therapeutic Guidelines (loading dose of 25 mg/kg followed by maintenance dose of 15-20 mg/kg every 12 hours) with subsequent adjustment to maintain trough levels at 15-20 mg/dL OR Intravenous daptomycin 6-10 mg/kg per day, adjusted for renal function (details of renally adjusted dosing provided in full protocol).
  The choice of daptomycin or vancomycin is clinician-determined and may be influenced by such factors as local practice, the vancomycin minimum inhibitory concentration (MIC) of the isolate and evidence emerging during the course of the study
- Standard therapy + Beta-Lactam (Experimental): In addition to standard treatment an intravenous Beta-Lactam (β-lactam) will be added for the first 7 calendar days following randomisation (randomisation is day 1 - hence patients will receive 6-7 days of β-lactam). This β-lactam will be intravenous flucloxacillin 2g every 6 hours in Australia and intravenous cloxacillin 2g every 6 hours in Singapore. For those with a history of minor allergy to any penicillin (rash or unclear history, but not anaphylaxis or angiooedema), it will be intravenous cefazolin 2g every 8 hours. For haemodialysis patients, it will usually be cefazolin 2g three times per week post dialysis, however clinicians are also free to choose intermittent (flu)cloxacillin, dosed as for glomerular filtration rate (GFR ) <10, if they desire.
  Interventions: Drug: Beta-Lactam

INTERVENTIONS:
Drug: Beta-Lactam
  Other Names: flucloxacillin; cloxacillin; cephazolin
  Arms: Standard therapy + Beta-Lactam

SUMMARY:
The aim of this clinical trial is to determine whether a novel combination antibiotic treatment (vancomycin/daptomycin + beta-lactam) is superior to the standard antibiotic treatment (vancomycin/daptomycin) for hospitalised adults with Methicillin Resistant Staphylococcus aureus bacteraemia. The hypothesis is that the addition of beta-lactam antibiotics (these are antibiotics from the penicillin family) to the standard therapy will lead to more efficient bacterial killing and hence lead to faster clearance of bacteria from the blood stream and other areas of infection, thereby reducing the risk of the spread of infection and death.

The study design is an investigator-initiated, multi-centre, open-label, randomised controlled trial. This will include 440 participants diagnosed with Methicillin Resistant Staphylococcus aureus bacteraemia recruited over a period of 4 years (July 2015 - June 2019) from within Infectious Diseases inpatient units across 21 hospital sites including 18 from within Australia and 3 located in Singapore. Participation will be voluntary and subject to informed consent. The participants will be randomised 1:1 to either the standard therapy group or combination therapy group. The combination therapy will include a treatment of intravenous beta-lactam for the first 7 days of treatment, in addition to the standard treatment (either vancomycin or daptomycin). The primary outcome measure will be complication-free survival 90 days post randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. ≥1 set of blood cultures positive for MRSA
3. Able to be randomized within 72 hours of blood cultures being collected.
4. Likely to remain as inpatient for 7 days following randomization

Exclusion Criteria:

1. Previous type 1 hypersensitivity reaction to ß-lactams
2. Polymicrobial bacteraemia (not counting contaminants)
3. Previous participation in the trial
4. Known pregnancy
5. Current β-lactam antibiotic therapy which cannot be ceased or substituted
6. Participant's primary clinician unwilling to enrol patient
7. Moribund (expected to die in next 48 hours with or without treatment)
8. Treatment limitations which preclude the use of antibiotics Note that we are NOT planning to exclude participants with renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Complication-free 90 day survival | Time period from randomisation (day 1) to day 90
  Composite outcome at 90 days - any of:
  1. All-cause mortality
  2. Persistent bacteraemia at day 5 or beyond
  3. Microbiological relapse - positive blood culture for MRSA at least 72 hours after a preceding negative culture
  4. Microbiological treatment failure. Positive sterile site culture for MRSA at least 14 days after randomisation.

SECONDARY OUTCOMES:
All-cause mortality at days 14, 42 and 90 days | Time period from randomisation (day 1) to day 90
Persistent bacteraemia at day 2 | Time period from randomisation (day 1) to day 90
Persistent bacteraemia at day 5 or beyond | Time period from randomisation (day 1) to day 90
Acute kidney injury defined as ≥ stage 1 modified RIFLE criteria at any time within the first 7 days, OR new need for renal replacement therapy at any time from days 1 to 90. Excludes participants already on haemodialysis. | Time period from randomisation (day 1) to day 90
  >=stage 1 modified RIFLE criteria (1.5-fold increase in the serum creatinine, or glomerular filtration rate (GFR) decrease by 25 percent). This endpoint does not apply to participants who were already on haemodialysis at randomisation.
Microbiological relapse - positive blood culture for MRSA at least 72 hours after a preceding negative culture | Time period from randomisation (day 1) to day 90
Microbiological treatment failure. Positive sterile site culture for MRSA at least 14 days after randomisation | Time period from randomisation (day 1) to day 90
Duration of intravenous antibiotic treatment | Time period from randomisation (day 1) to day 90
Direct health care costs | Time period from randomisation (day 1) to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Davis, MBBS, FRACP, Principal Investigator — Menzies School of Health Research; Steven Tong, MBBS, FRACP, Principal Investigator — Menzies School of Health Research
Locations (30):
- Australia (24):
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Darwin Hospital, Darwin, Northern Territory
  - Cairns Hospital, Cairns, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinder's Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Medical Centre Clayton Campus, Clayton, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - Western Health - Footscray, Footscray, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Western Health - Sunshine Hospital, Sunshine, Victoria
  - Western Health - Williamstown Hospital, Williamstown, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Israel (2):
  - Rambam Health Corporation, Haifa
  - Beilinson Hospital, Petah Tikva
- Middlemore Hospital, Otahuhu, Auckland, New Zealand
- Singapore (3):
  - Tan Tock Seng Hospital, Novena, Tan Tock Seng
  - National University Hospital, Kent Ridge
  - Singapore General Hospital, Outram Park

REFERENCES:
- [Derived] Tong SYC, Lye DC, Yahav D, Sud A, Robinson JO, Nelson J, Archuleta S, Roberts MA, Cass A, Paterson DL, Foo H, Paul M, Guy SD, Tramontana AR, Walls GB, McBride S, Bak N, Ghosh N, Rogers BA, Ralph AP, Davies J, Ferguson PE, Dotel R, McKew GL, Gray TJ, Holmes NE, Smith S, Warner MS, Kalimuddin S, Young BE, Runnegar N, Andresen DN, Anagnostou NA, Johnson SA, Chatfield MD, Cheng AC, Fowler VG Jr, Howden BP, Meagher N, Price DJ, van Hal SJ, O'Sullivan MVN, Davis JS; Australasian Society for Infectious Diseases Clinical Research Network. Effect of Vancomycin or Daptomycin With vs Without an Antistaphylococcal beta-Lactam on Mortality, Bacteremia, Relapse, or Treatment Failure in Patients With MRSA Bacteremia: A Randomized Clinical Trial. JAMA. 2020 Feb 11;323(6):527-537. doi: 10.1001/jama.2020.0103. PMID 32044943
- [Derived] Tong SY, Nelson J, Paterson DL, Fowler VG Jr, Howden BP, Cheng AC, Chatfield M, Lipman J, Van Hal S, O'Sullivan M, Robinson JO, Yahav D, Lye D, Davis JS; CAMERA2 study group and the Australasian Society for Infectious Diseases Clinical Research Network. CAMERA2 - combination antibiotic therapy for methicillin-resistant Staphylococcus aureus infection: study protocol for a randomised controlled trial. Trials. 2016 Mar 31;17:170. doi: 10.1186/s13063-016-1295-3. PMID 27029920